CLINICAL TRIAL: NCT07083674
Title: TeamTalk: Strategies to Improve Communication Structure and Quality in Low-resource Childhood Cancer Hospitals
Brief Title: TeamTalk: Improving Inter-professional Communication During Cancer Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: St. Jude Children's Research Hospital (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sara Malone, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202503183; 1R01CA287374 (NIH)
Record Dates: First submitted 2025-07-08; First posted 2025-07-24 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Cancer
Keywords: Pediatric Cancer; Communication
MeSH Terms: conditions — Neoplasms; Communication

STUDY DESIGN:
Intervention Model Description: Parallel-arm, pilot cluster-randomized wait list-controlled trial to evaluate the intervention compared to control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This study includes an intervention development phase (Aim 2) during which the intervention content and delivery mechanisms will be finalized. We will implement the multilevel intervention developed in Aim 2. We anticipate this will consist of one instance of intervention at each hospital and we will develop a full intervention manual following Aim 2. Details regarding the intervention will be updated prior to participant enrollment in the trial.
  Interventions: Behavioral: Multi-level communication intervention
- Waitlist Control Group (No Intervention): The wait list control is a group that does not receive an intervention during the study period, serving as an untreated comparison during the study, although they later receive the intervention. This intervention will be delivered after the completion of the last data collection instance.

INTERVENTIONS:
Behavioral: Multi-level communication intervention — The intervention will target multiple levels (provider, unit, hospital) and will respond to identified modifiable communication challenges. Aim 2 intervention mapping will finalize the specific intervention; we anticipate it will involve training and education of staff members and new unit protocols for communication.
  Arms: Intervention Group

SUMMARY:
This study focuses on improving interprofessional communication during cancer treatment, through an individual and hospital system intervention, to improve provider outcomes, patient care, and, ultimately, survival for children with cancer in low-resource settings.

ELIGIBILITY:
Inclusion Criteria:

* Hospitals identified as being in lowest quartile of communication quality, as defined by prior cross-sectional CritCom analysis and measured as the overall CritCom score.
* All Global Alliance hospitals providing childhood cancer care will be eligible to participate.
* Individual participants will be included if they care for hospitalized children with cancer at risk of deterioration.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2027-09-23 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Communication quality - CritCom Measure | We will evaluate outcomes at three time points; baseline, one month after intervention, and six months after intervention.
  Reliable, published measure of communication quality; measured across 6 domains on a Likert scale; self reported by clinical team members; Will assess change in clinician perspective of communication quality within 6 months

OTHER OUTCOMES:
Provider burnout and retention | We will evaluate outcomes at three time points; baseline, one month after intervention, and six months after intervention.
  Provider outcomes will be assessed at the individual level via questions about burnout and intent to leave. This will use pre-existing, reliable measures where individuals report their self-reported rates of burnout and intent to leave their job. These are categorical responses.
Patient mortality and safety/adverse events | We will evaluate outcomes at three time points; baseline, one month after intervention, and six months after intervention.
  Patient outcomes data will be collected via prospective registry of all clinical deterioration events, defined as unplanned transfers to intensive care (ICU), the use of ICU interventions on general wards, or unplanned death on the ward.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DEVELOPMENT OF A QUANTITATIVE MEASURE (CRITCOM) TO ASSESS THE QUALITY OF INTERDISCIPLINARY COMMUNICATION AROUND PATIENT DETERIORATION IN VARIABLY RESOURCED HOSPITALS
- [Derived] Agulnik A, Graetz DE, Carothers BJ, Rivera J, Blakeney EA, Hayes S, Chaitan VL, Cabassa L, Goss CW, Luke DA, Malone S. Strategies to improve healthcare team communication structure and quality in resource-variable childhood cancer hospitals (TeamTalk): a study protocol. Implement Sci Commun. 2025 Nov 17;6(1):124. doi: 10.1186/s43058-025-00811-z. PMID 41250257